CLINICAL TRIAL: NCT00729300
Title: Laboratory Models of Cocaine Self-administration
Brief Title: A Study of the Relationship Between Disulfiram and Cocaine Self-administration.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Christopher Verrico, Associate Professor, Psychiatry Research, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-23131
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Cocaine Addiction
Keywords: cocaine; disulfiram; antabuse; addiction; stimulant
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Disulfiram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 2 (Experimental): disulfiram
  Interventions: Drug: disulfiram

INTERVENTIONS:
Drug: placebo — 0mg daily
  Arms: 1
Drug: disulfiram — 250mg daily
  Arms: 2

SUMMARY:
The problem of cocaine dependence remains a major medical, social, and legal concern. Several studies have suggested that disulfiram may be beneficial for the treatment of cocaine dependence. A common assumption has been that disulfiram treatment, by increasing DA availability, enhances the aversive aspects of stimulants. This study aims to measure plasma activity in those with the C/C DBH genotype, which is associated with higher DBH activity subsequently making the disulfiram treatment more effective, as well as determine the effects of treatment with disulfiram on cocaine self-administration using a human laboratory model of cocaine self-administration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meet DSM IV criteria for cocaine dependence; 2. Have a self-reported history of using cocaine by the smoked or IV route. Participants must report at least weekly use for the past month and have a cocaine-positive urine test in the week of study entry; 3. Have vital signs after a 48 hours washout period as follows: resting pulse between 50 and 80 bpm, blood pressures between 105-130mm Hg systolic and 45-80mm Hg diastolic; 4. Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal; 5. Have a baseline ECG that demonstrates normal sinus rhythm, normal conduction, and no clinically significant arrhythmias; and 6. Have a medical history and standard physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.

Exclusion Criteria:

* 1. Have any history or evidence suggestive of seizures or brain injury 2. Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, or epileptic seizure; 3. Have neurological or psychiatric disorders, such as:

  * psychosis, bipolar illness or major depression as assessed by MINI (or SCID if necessary);
  * organic brain disease or dementia assessed by clinical interview;
  * history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult;
  * history of suicide attempts within the past three months assessed by MINI and/or current suicidal ideation/plan as assessed by MINI; 4. Have evidence of clinically significant heart disease or hypertension, as determined by the PI; 5. Have a family history in first degree relatives of early cardiovascular morbidity or mortality, as determined by the PI; 6. Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease; 7. Have HIV and are currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication; 8. Have any history of asthma, chronic coughing and wheezing, or other respiratory illnesses; 9. Heavy current alcohol intake that is likely to lead to withdrawal symptoms, in the opinion of the PI; 10. Refuse to abstain from alcohol during the protocol and for at least one week after discharge.

    11. Have any other illness, condition, or use of medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2006-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, MD, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haile CN, De La Garza R 2nd, Mahoney JJ 3rd, Nielsen DA, Kosten TR, Newton TF. The impact of disulfiram treatment on the reinforcing effects of cocaine: a randomized clinical trial. PLoS One. 2012;7(11):e47702. doi: 10.1371/journal.pone.0047702. Epub 2012 Nov 8. PMID 23144826

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  placebo: placebo daily
- Disulfiram Treatment Group: disulfiram
  disulfiram: 250mg daily
Period: Overall Study
Arm/Group | Placebo | Disulfiram Treatment Group
Started | 26 | 26
Completed | 17 | 17
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Population: Only data from study completers was considered
Groups:
- Placebo Group: Placebo
  placebo: placebo daily
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Disulfiram Treatment Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.41 (1.61) | 41.41 (1.61) | 41.41 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 15 | 15 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Self-administration
Description: The reinforcing effects of cocaine were determined using a self-administration procedure in which subjects choose to take previously sampled doses of cocaine or cash of increasing monetary value. The mean number of cocaine choices across each drug condition (i.e., placebo and disulfiram) is reported.
Time Frame: 4 days
Population: Only data from study completers was considered
Measure: Mean (Standard Error); unit: cocaine choices/participant
Units Other Than Participants: cocaine choices
Arm/Group | Placebo | Disulfiram Treatment Group
Number analyzed (Participants) | 17 | 17
Number analyzed (cocaine choices) | 170 | 170
cocaine choices/participant | 2.5 (0.5) | 4.8 (0.8)

ADVERSE EVENTS:
Groups:
- Disulfiram: disulfiram
  disulfiram: 250mg daily
Arm/Group | Placebo | Disulfiram
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
First, we focused on behavioral effects and did not obtain subjective measures (i.e., euphoria and craving). This could have contributed to our understanding of how disulfiram enhanced cocaine's reinforcing effects. Second, we administered cocaine by the IV route whereas a majority of our participants took cocaine by smoking, and this may have influenced certain outcomes. Finally, we treated participants for only a few days, whereas clinical trials last much longer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No